CLINICAL TRIAL: NCT01695967
Title: Turbinate Cauterization in Pediatric Patients With Nasal Obstruction A Randomized Prospective Trial
Brief Title: Turbinate Cauterization in Pediatric Patients With Nasal Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Responsible Party: Principal Investigator, Cristina Baldassari M.D., Assistant Professor, Pediatric Otolaryngology, Eastern Virginia Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: version 3 03Mar2012
Record Dates: First submitted 2012-09-24; First posted 2012-09-28 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Sleep Apnea; Nasal Obstruction
Keywords: nasal obstruction
MeSH Terms: conditions — Sleep Apnea Syndromes; Nasal Obstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Turbinate Cauterization (Experimental): Turbinate Cauterization will be completed.
  Interventions: Procedure: turbinate cauterization
- control (No Intervention): no turbinate cauterization

INTERVENTIONS:
Procedure: turbinate cauterization
  Arms: Turbinate Cauterization

SUMMARY:
patients will be placed in 2 groups, with or without turbinate cautery ( a surgical method to reduce the size of the skin covered bones in the nose), at the time of adenoidectomy and tonsillectomy. It will compare the amount of nasal congestion for each group with the idea that it will be less if treated with turbinate cauterization. Assessments from baseline to 6 months post procedure will be compared between the two groups.

DETAILED DESCRIPTION:
To assess if inferior turbinate cautery improves nasal obstruction in children undergoing adenotonsillectomy.

ELIGIBILITY:
Inclusion Criteria:

* ages 3-16
* obstructive sleep apnea warranting adenotonsillectomy
* history of daytime nasal obstruction and or mouth breathing
* failed medical treatment with either oral anti-histamine or nasal steroid spray.
* turbinate hypertrophy on Physical Exam defined by >50% obstruction

Exclusion Criteria:

* <3 or >16
* unwillingness to comply with study procedures
* congenital head and neck malformations, genetic syndromes, craniofacial anomalies
* no evidence of turbinate hypertrophy or symptoms of nasal obstruction
* pregnancy or breastfeeding
* bleeding disorders
* current therapy with coumadin or Pradaxa

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2012-08 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
# of participants with improved nasal obstruction score from baseline to 6 months | baseline and 6 months
  Baseline assessment compared to 6 mo post surgery. The SN-5 Nasal Obstruction and Sinonasal Quality of Life instrument tools will be used to record nasal obstruction symptom scores.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Baldassari, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Children's Hospital of the King's Daughters, Norfolk, Virginia, United States